CLINICAL TRIAL: NCT03771443
Title: Assessment of the Effect of Gluten Free Toothpaste on the Ulcerative Events in Children With Celiac Disease (Before and After Pilot Study)
Brief Title: Assessment of the Effect of Gluten Free Toothpaste on the Ulcerative Events in Children With Celiac Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Adel Abd Elhameed, master degree student, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-12-01
Record Dates: First submitted 2018-12-08; First posted 2018-12-11 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Gluten Sensitivity
Keywords: Gluten-free toothpaste,celiac disease, GFD, children
MeSH Terms: conditions — Celiac Disease; Jones syndrome | interventions — green tea bioflavonoid, zinc ascorbate-containing toothpaste

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gluten free toothpaste (Experimental): experimental gluten free toothpaste with natural ingredients prepared for the study to be used 3 times per day for six months
  Interventions: Drug: experimental gluten free toothpaste

INTERVENTIONS:
Drug: experimental gluten free toothpaste — we prepared gluten free toothpaste in the faculty of pharmacy -Cairo university because there is no gluten free toothpaste available in the Egyptian market .
  Other Names: natural toothpaste

SUMMARY:
Celiac disease (CD) is the most common genetically based food intolerance in the world, with a prevalence among approximately 1% of the general population (Guandalini & Assiri, 2014). CD is a frequent disorder among Egyptian children, both in the general population and in at-risk groups(Abu-Zekry et al., 2008). It is estimated that the incidence of CD is 3 to13 cases per1000, with a higher prevalence among first-degree relatives of patients with CD.Lifelong adherence to a strict gluten free diet (GFD) remains the only available treatment for patients with CD and typically results in a complete return to health. Nevertheless, gluten is not found only in diet, Gluten is commonly used as a binder in products like medication, cosmetics, oral and skin care, and even children's toys. Gluten is found also in toothpastes and other oral health products and it can be swallowed by mistake and initiate immune response(Anon, n.d.). Unfortunately, there is no gluten free toothpaste available in the Egyptian market and it is very expensive if we bought it from Europe or USA. The tube will cost nearly 10 dolars .As a result, the production and availability of gluten free toothpaste in Egypt has become mandatory.

DETAILED DESCRIPTION:
production of an experimental gluten free toothpaste and providing it for children with celiac disease

ELIGIBILITY:
Inclusion Criteria:

1. Age above 6 yeas.
2. Erupting lower 6.
3. Can spit the toothpaste.
4. Diagnosed as a celiac patient(pathology&serology)

Exclusion Criteria:

1. With a history of allergy to any ingredient present in the toothpaste to be used for treatment
2. The presence of serious medical conditions or a transmissible disease such as malignant disease, hepatitis, AIDS etc.
3. Children whose parents had no home or mobile phone to enable post-operative contact.
4. Parent that will not sign the consent.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-07-21 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Ulcerative events | Six months
  Reporting from the parent (Yes or No)

SECONDARY OUTCOMES:
Inflammation or ulceration | six months
  visual (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Abdelhameed, BSc, Principal Investigator — Resident at Pediatric Dentistry and Dental Public Health Department; Fatma KI Abdelgawad, PhD, Study Chair — Assistant Professor at Pediatric Dentistry and Dental Public Health Department; Kamal M El Motayam, PhD, Study Director — Emeritus Professor at Pediatric Dentistry and Dental Public Health Department
Locations (1):
- Faculty of Dentistry, Cairo University, Giza, Al Manial, Cairo, Egypt, Egypt